CLINICAL TRIAL: NCT02236494
Title: Pilot Trial of Emergency Department Intervention and Referral for Alcohol Misuse in Older Adults
Brief Title: Study of an Emergency Department-based Intervention to Reduce Alcohol Misuse in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: The American Geriatrics Society (Other); National Institute on Aging (NIA) (NIH); Society for Academic Emergency Medicine (Other); North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13-3446; R03AG048090 (NIH)
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Alcohol Abuse
Keywords: alcoholism; dangerous behavior; aged; emergency medicine
MeSH Terms: conditions — Alcoholism; Dangerous Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- General Health Information Pamphlet (Active Comparator): This group will not receive a brief intervention in the ED. They will receive a pamphlet with general health information for older adults, as well as contact information for an outpatient alcohol treatment center where they have the option to follow-up for alcohol treatment at their discretion. The patient's readiness to change their alcohol habits will be measured using a 1-10 scale with a visual cue.
  Interventions: Behavioral: General Health Information
- Brief Negotiated Interview (Experimental): The BNI will follow standard steps (7, 63): 1. The research assistant (RA) will ask permission to discuss the patient's alcohol use with them. 2. They will provide feedback regarding the patient's alcohol use, and will review guidelines drinking in older adults. Where relevant, the RA will discuss how the patient's current visit may relate to their alcohol use. 3. The RA will assess the patient's readiness to change using a 1-10 scale, and will enhance motivation. 4. The RA will negotiate a goal for the patient's drinking and give advice. The patient will be asked to sign a drinking agreement.
  Interventions: Behavioral: Brief Negotiated Interview

INTERVENTIONS:
Behavioral: Brief Negotiated Interview — As per arm
  Arms: Brief Negotiated Interview
Behavioral: General Health Information — As per arm (this is the active comparator)
  Arms: General Health Information Pamphlet

SUMMARY:
This is a randomized trial to assess the value of an emergency department-based intervention to reduce hazardous alcohol use among older adults. We hypothesize that the intervention will result in a 25% reduction in the prevalence of hazardous alcohol use while the control group will only have a 5% reduction.

DETAILED DESCRIPTION:
The goal of this project is to perform a pilot, randomized, controlled trial of a brief intervention and referral for treatment among older adults in the emergency department (ED) with alcohol misuse. The pilot data would then be used to design a larger study. The intervention for this trial will consist of a Brief Negotiation Interview (BNI) with a stratified referral for further treatment, compared with usual care. The BNI is a standardized, well-described intervention that has been implemented in a broad range of clinical settings but has not been specifically tested in older adults in the ED. Following the BNI, we will provide a referral for further care for the patient that is stratified by severity of alcohol misuse. Patients with hazardous or harmful alcohol use will follow-up with a primary care physician; patients with alcohol abuse or dependence will follow-up with an outpatient alcohol and substance abuse program; those at risk for complicated withdrawal will be recommended for inpatient treatment. In all cases we will contact the referral physician to help transition the patient's care, and ensure the patient receives a consistent message regarding their alcohol use across the different care settings.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 and older
* Receiving care in the emergency department
* Hazardous alcohol use, defined as reporting drinking more than 7 drinks per week on an average week during the three months prior to the visit, and whether they have consumed more than three drinks on any given occasion.

Exclusion Criteria:

* Prisoner
* psychosis or psychiatric hold
* nursing home
* life-threatening condition
* current hospice care

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 222 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-07-10 (Actual); Study Completion 2017-07-10 (Actual)

PRIMARY OUTCOMES:
Alcohol misuse | 6 months
  Self-reported alcohol misuse is defined as patient self-report of either drinking >7 drinks per week or >3 drinks per occasion in the past month.
Subgroup analysis of patients who met hazardous alcohol use criteria based on time-line follow back method of assessing alcohol consumption | 6 months
  Analysis of rate of hazardous alcohol use in the control and intervention arms within the subgroup of patients who met hazardous drinking criteria of >7 drinks in the past 7 days, or >3 drinks per occasion within the last 28 days using the time-line follow back method.

SECONDARY OUTCOMES:
Alcohol misuse | 3 months, 12 months
  Alcohol misuse is defined as patient self-report of either drinking >7 drinks per week or >3 drinks per day in the past month.
Function | 6,12 months
  Activities of Daily Living
Alcohol consumption | 3,6,12 months
  Average drinks per week and episodes of >3 drinks in past 3 months
Alcohol abuse | 3,6,12 months
  AUDIT Score
General Health | 3,6,12 months
  Mobility, depression, and presence of chronic pain
Risk-taking behavior | 6,12 months
  Driving after drinking
Trauma | 6,12 months
  Injuries, falls, and motor vehicle collisions within the last 6 months, alcohol use preceding and medical care following the injury
Healthcare Utilization | 6,12 months
  Number of primary care, urgent care, and ED visits, and hospitalization days within the last 6 months, and any relation of these visits to alcohol use.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Shenvi, MD,PhD, Principal Investigator — UNC Chapel Hill; Timothy F Platts-Mills, MD,MSc, Principal Investigator — UNC Chapel Hill
Locations (1):
- UNC Hospitals Emergency Department, Chapel Hill, North Carolina, United States